CLINICAL TRIAL: NCT07405931
Title: Evaluation of the Effectiveness of Managing Chemotherapy Side Effects Using ePRO and a Standardized Telenursing Program for Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government); Kosin University Gospel Hospital (Other); Gyeongsang National University Hospital (Other); Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Koh Su-Jin, Professor, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-05-022
Record Dates: First submitted 2026-01-22; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Early Gastric Cancer; Advanced Gastric Cancer; Early Lung Cancer; Advanced Lung Cancer; Early Breast Cancer; Advanced Breast Cancer; Early Colon Cancer; Advanced Colon Cancer
MeSH Terms: conditions — Stomach Neoplasms; Lung Neoplasms; Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care Group (No Intervention): Standard care group is the control group, receiving standard care only without using Smart Cancer Care Plus or standardized telenursing.
- ePRO Group (Experimental): ePRO group is the experimental group, using Smart Cancer Care Plus without standardized telenursing.
  Interventions: Other: Smart Cancer Care Plus
- ePRO + Telenursing Group (Experimental): ePRO + Telenursing group is the experimental group, using Smart Cancer Care Plus in combination with standardized telenursing.
  Interventions: Other: Standardized Telenursing; Other: Smart Cancer Care Plus

INTERVENTIONS:
Other: Standardized Telenursing — Within Smart Cancer Care Plus, predefined criteria are applied to trigger standardized telenursing interventions. When patients report symptoms of Grade 3 or higher severity, or when a scheduled weekly symptom report is not submitted within 48 hours of the designated reporting date, a structured telephone counseling session is initiated. This process is intended to ensure timely clinical follow-up, support appropriate self-management, and prevent the progression of unmanaged adverse events.
  Arms: ePRO + Telenursing Group
Other: Smart Cancer Care Plus — Smart Cancer Care Plus is a digital platform for patient-reported symptom monitoring and management, developed for individuals receiving chemotherapy. The system enables structured reporting of chemotherapy-related adverse events and provides standardized information regarding the severity grading of symptoms, accompanied by evidence-based self-management strategies. This intervention is intended to promote systematic symptom monitoring and to facilitate timely clinical responses to adverse events.
  Other Names: Smart Caner Care Plus
  Arms: ePRO + Telenursing Group; ePRO Group

SUMMARY:
This is a multicenter randomized controlled clinical trial designed to evaluate the clinical efficacy and cost-effectiveness of a digital health platform that integrates a symptom reporting and management software with a standardized telenursing program, allowing cancer patients to actively monitor, report, and self-manage chemotherapy-related adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Diagnosed with early or advanced gastric, lung, breast, or colon cancer
* Starting first-cycle chemotherapy with a new anticancer agent
* Able to use a smartphone without difficulty
* Willing to provide informed consent to participate in the study

Exclusion Criteria:

* Individuals who have difficulty communicating due to cognitive impairment, visual impairment, hearing impairment, or other reasons
* Individuals who cannot read, write, or understand Korean
* Other individuals deemed inappropriate for participation by the investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life Measured by EORTC QLQ-C30 | 12 weeks
  Quality of life will be assessed using the Global Health Status/Quality of Life scale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). The score for the Global Health Status/Quality of Life scale ranges from 0 to 100, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Self-management, which will be assessed using the SECD-6-K | 6 months
  Self-management will be assessed using the Self-Efficacy for Chronic Disease Scale-6 Item, Korean Version (SECD-6-K). The SECD-6-K consists of 6 items, each rated on a 10-point Likert scale (1-10). The total score ranges from 6 to 60, with higher scores indicating better self-management.
Self-rated overall health, which will be assessed using EQ-5D-VAS | 6 months
  Self-rated overall health will be assessed using the EuroQol Visual Analogue Scale (EQ-5D-VAS). Participants rate their overall health on a visual analogue scale ranging from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. Higher scores indicate better self-rated health.
Adherence to ePROSW | 6 months
  Adherence to ePROSW will be assessed by measuring the frequency of app usage over the entire 6-month study period. App adherence is defined as the total number of times participants accessed and used the ePROSW application during the study period.
Chemotherapy Adherence | 6 months
  Chemotherapy adherence will be evaluated by the percentage of planned chemotherapy completed. Adherence will be calculated as the ratio of the administered dose to the planned dose, expressed as a percentage.
Healthcare Utilization | 6 months
  Healthcare utilization will be assessed by the occurrence of unplanned hospital visits during the study period.
Functional status, which will be assessed using EORTC-QLQ-C30 | 6 months
  Functional status will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). The functional scales include physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning. Scores for each scale are linearly transformed to a 0-100 scale, with higher scores indicating better functioning.
Symptom severity, which will be assessed using EORTC-QLQ-C30 | 6 months
  Symptom severity will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). The symptom scales include fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties. Scores for each symptom scale are linearly transformed to a 0-100 scale, with higher scores indicating greater symptom severity (worse outcome).
Satisfaction, which will be assessed using system usability scale | 6 months
  User satisfaction with the system will be assessed using the System Usability Scale (SUS), a validated 10-item questionnaire. Each item is rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). The total SUS score is calculated by multiplying the sum of item scores by 2.5, resulting in a range of 0 to 100, where higher scores indicate greater satisfaction (better usability).

CONTACTS AND LOCATIONS:
Overall Officials: Sujin Koh, Doctor of Philoshophy, Principal Investigator — Ulsan University Hospital; Keun Soek Lee, Doctor of Philoshophy, Principal Investigator — National Cancer Center, Korea; Sung Hoon Sim, Doctor of Philoshophy, Principal Investigator — National Cancer Center, Korea; Ji Hyung Hong, Doctor of Philoshophy, Principal Investigator — National Cancer Center, Korea; Sun Jin Sym, Doctor of Philoshophy, Principal Investigator — Gachon University Gil Medical Center; Jung Hun Kang, Doctor of Philoshophy, Principal Investigator — Gyeongsang National University Hospital; Seong Hoon Shin, Doctor of Philoshophy, Principal Investigator — Kosin University Gospel Hospital
Locations (5):
- South Korea (5):
  - Kosin University Gospel Hospital, Busan
  - National Cancer Center, Korea, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University, Jinju
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF